CLINICAL TRIAL: NCT01702766
Title: Bifidobacterium Animalis Subsp. Lactis for Lowering the Risk of Common Infections in Hospitalized Children
Acronym: PROBIC II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Zagreb (Other)
Responsible Party: Sponsor
Model: Parallel | Purpose: Prevention
Other Study IDs: PROBBIC II Study
Record Dates: First submitted 2012-10-03; First posted 2012-10-08 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Gastrointestinal Tract Infections; Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bifidobacterium animalis subsp. lactis (Active Comparator)
  Interventions: Dietary Supplement: Bifidobacterium animalis subsp. lactis
- Placebo (Placebo Comparator)

INTERVENTIONS:
Dietary Supplement: Bifidobacterium animalis subsp. lactis
  Arms: Bifidobacterium animalis subsp. lactis

SUMMARY:
Hypothesis: Use of Bifidobacterium animalis subsp. lactis can effectively prevent common nosocomial (gastrointestinal and respiratory) infections. Nosocomial infection will be defined as infections which develop more than 48 hours after admission and they are not present or incubating on admission

This study is a prospective, randomized, double blind, placebo- controlled parallel study in children hospitalized at Children's hospital Zagreb.

The study will investigate the effect of supplementation with the probiotic strain Bifidobacterium animalis subsp. lactis on the incidence and duration of gastrointestinal and respiratory infections.

The test product is a sachet containing 1 gram of powder. The test product will contain minimum 1 billion CFU (colony forming units) probiotic per serving.

The placebo product is an identical product except for the absence of probiotics.

The study includes an intervention period lasting the length of the hospital stay.

The study product will be consumed daily in the morning together with breakfast.

The consumption of the study products will be taken under the surveillance of the physician.

Data on infections will be diagnosed by a physician and recorded in a CRF. The incidence of infections will be analyzed based on the information recorded in the CRF.

ELIGIBILITY:
Inclusion Criteria:

* Children hospitalized at the Department of Paediatrics, Children's Hospital Zagreb
* Age from 1 year to 18 years
* Signed informed consent by the parents

Exclusion Criteria:

* Immunodeficiency
* Infants from neonatal period until 1 year of age
* Re-hospitalisation (readmission in a hospital within one month)
* Receiving probiotic and /or prebiotic products prior to enrolment (2 weeks prior to hospitalization)
* Neoplasms
* Severe chronic diseases
* Hospitalization shorter than 3 days

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Dates: Start 2012-12; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Common infections in children
  Number of children with common infections (gastrointestinal and respiratory infections):
  Gastrointestinal tract infections defined as diarrhoea (3 or more loose or watery stools in 24 hours or increase of number of stools for more than 50% in 24 hours) or vomiting (defined by physician and not a result of other symptoms including cough or diseases including gastroesophageal reflux disease or neurological conditions) or both.
  Respiratory tract infections defined as: pharyngitis, otitis, common cold, pneumonia, bronchitis and bronciolitis (all infections diagnosed by physician) Number of children with adverse events.

SECONDARY OUTCOMES:
Duration of symptoms
  Duration of symptoms in days

OTHER OUTCOMES:
Severity of infection
  Severity of GI infections based on Vesikari scale Severity of respiratory infections according to the physician based on visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Zagreb, Zagreb, Croatia

REFERENCES:
- [Derived] Hojsak I, Tokic Pivac V, Mocic Pavic A, Pasini AM, Kolacek S. Bifidobacterium animalis subsp. lactis fails to prevent common infections in hospitalized children: a randomized, double-blind, placebo-controlled study. Am J Clin Nutr. 2015 Mar;101(3):680-4. doi: 10.3945/ajcn.114.102004. Epub 2015 Jan 7. PMID 25733653